CLINICAL TRIAL: NCT01683396
Title: A Phase 2 Proof-of-Concept Study of Gevokizumab in Active Inflammatory, Erosive Osteoarthritis of the Hand
Brief Title: Safety and Biologic Activity Study of Gevokizumab to Treat Erosive Osteoarthritis of the Hand
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: X052160
Record Dates: First submitted 2012-09-06; First posted 2012-09-11 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthritis
Keywords: Erosive Osteoarthritis; Osteoarthritis; Osteoarthritis of the Hand
MeSH Terms: conditions — Osteoarthritis | interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- gevokizumab (Experimental)
  Interventions: Drug: gevokizumab

INTERVENTIONS:
Drug: Placebo — Solution for subcutaneous injection
  Arms: Placebo
Drug: gevokizumab — Solution for subcutaneous injection
  Arms: gevokizumab

SUMMARY:
The purpose of this proof-of-concept study is to determine whether gevokizumab is effective in the treatment of active inflammatory, erosive osteoarthritis of the hand.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hand osteoarthritis
* Joint tenderness and/or redness
* At least one erosion by X-ray (as determined by the central reader)
* Contraceptive measures adequate to prevent pregnancy during the study

Exclusion Criteria:

* History of inflammatory disease other than hand EOA including: secondary post-traumatic OA; rheumatoid arthritis; spondylarthropathies; erosion of the ulnar styloid process; psoriatic arthritis; skin psoriasis; erosions of the wrist; fibromyalgia
* History of gout, pseudogout, or hemochromatosis
* History of allergic or anaphylactic reactions to monoclonal antibodies
* History of recurrent or chronic systemic infections
* Known allergy to acetaminophen
* Female subjects who are pregnant, planning to become pregnant, have recently delivered, or are breast-feeding

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in AUSCAN pain score at Day 84 | Baseline and Day 84
  The Australian/Canadian (AUSCAN) Osteoarthritis Hand Index is a self-report assessment of pain, stiffness, and function in patients with hand osteoarthritis.

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Huntsville, Alabama
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Roseville, California
  - Sacramento, California
  - Santa Monica, California
  - Van Nuys, California
  - Denver, Colorado
  - Miami, Florida
  - Pinellas Park, Florida
  - Sarasota, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Wichita, Kansas
  - Reno, Nevada
  - New York, New York
  - Rochester, New York
  - Raleigh, North Carolina
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Waco, Texas
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Franklin, Wisconsin